CLINICAL TRIAL: NCT04630236
Title: Ultrasound Guided Positioning of Central Venous Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Collaborators: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CVC061120
Record Dates: First submitted 2020-11-06; First posted 2020-11-16 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Central Venous Catheter
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound (Other)
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Using ultrasound control, the central vein catheter is injected with saline solution and the time to detect the saline bolus in the ultrasound is measured.

SUMMARY:
The current standard for (correct) position control of a central venous catheter (CVC) is X-ray control, which is associated with X-rays for the patient. In some clinics, radiological services are not offered "around the clock". Therefore, an alternative that is not burdensome for patients and is available on all sides would be desirable. The possibility of a sonographic CVC position control is to be investigated.

The correct position of a central venous catheter is important. Complications/failure must be detected early/immediately. In addition to the X-ray of the thorax, a position control by means of an ECG derivative (α-card derivative) is available for position control. The method is easy to perform, but an epicardial or an arterial position of the CVC cannot be detected without the use of additional imaging in case of doubt.

For the reasons mentioned above, sonography is a suitable method to show the inflow of injected 0.9% sodium chloride solution into the right atrium, which allows to conclude the correct position of the CVC.

ELIGIBILITY:
Inclusion Criteria:

* elective insertion of a central venous catheter.

Exclusion Criteria:

* emergency insertion of a central venous catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
- correlation between the time of detection of the injected saline bolus and radiological position of the central venous catheter | up to 5 seconds
  - ultrasound during injection of saline solution into a newly inserted central venous catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologische Klinik Bad Salzhausen, Nidda, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schummer W, Schummer C, Schelenz C, Brandes H, Stock U, Muller T, Leder U, Huttemann E. Central venous catheters--the inability of 'intra-atrial ECG' to prove adequate positioning. Br J Anaesth. 2004 Aug;93(2):193-8. doi: 10.1093/bja/aeh191. Epub 2004 Jun 25. PMID 15220179
- [Background] Schummer W, Herrmann S, Schummer C, Funke F, Steenbeck J, Fuchs J, Uhlig T, Reinhart K. Intra-atrial ECG is not a reliable method for positioning left internal jugular vein catheters. Br J Anaesth. 2003 Oct;91(4):481-6. doi: 10.1093/bja/aeg208. PMID 14504146